CLINICAL TRIAL: NCT03745404
Title: A Double-blind, Multicentre, Multiple-dose, Enriched Enrolment, Randomized-withdrawal, Parallel-group Phase III Study With Lido-Patch and Corresponding Placebo Plaster in Patients Suffering From Postherpetic Neuralgia (PHN)
Brief Title: A Study With Lido-Patch and Placebo Plaster in Patients Suffering From Postherpetic Neuralgia (PHN)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Grünenthal GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: KF10004/01
Record Dates: First submitted 2018-11-15; First posted 2018-11-19 (Actual); Last update posted 2023-09-13 (Actual); Status verified 2023-09

CONDITIONS: Post Herpetic Neuralgia
Keywords: Post herpetic neuralgia; Lidocaine; Herpes zoster
MeSH Terms: conditions — Neuralgia, Postherpetic; Herpes Zoster | interventions — Lidocaine; Lidoderm

STUDY DESIGN:
Intervention Model Description: An enriched enrolment, randomized-withdrawal, parallel-group design was applied. Only participants responding to open-label active treatment were included into the Double-blind Phase.
  The study comprised:
  * A non-controlled, open-label enrichment phase with Lido-Patch treatment (Run-in Phase).
  * A double-blind, randomized-withdrawal phase (Double-blind Phase).
  * Upon request of the participant, treatment could be continued in the clinical study KF10004/02.
  * A Follow-up Phase without treatment for participants not continuing in KF10004/02.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Open-label enriched enrolment followed by double-blind treatment for 2 weeks.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Lido-Patch (Open-label Run-in Phase) (Experimental): All participants applied up to 3 Lido-Patches (lidocaine 5% medicated plaster) per day (depending on the size of PHN area). Patches were applied topically for up to 12 hours per day (patch free interval: at least 12 hours) at the site of skin affected by painful PHN.
  Interventions: Drug: Lidocaine 5% medicated Plaster
- Lido-Patch (Double-blind Phase) (Experimental): Up to 3 patches (lidocaine 5% medicated plaster) per day (depending on the size of PHN area) were applied topically for up to 12 hours per day (patch free interval: at least 12 hours) at the site of skin affected by painful PHN.
  Interventions: Drug: Lidocaine 5% medicated Plaster
- Placebo Patch (Double-blind Phase) (Placebo Comparator): Up to 3 placebo plasters per day (depending on the size of PHN area) were applied topically for up to 12 hours per day (patch free interval: at least 12 hours) at the site of skin affected by painful PHN.
  Interventions: Drug: Placebo Plaster

INTERVENTIONS:
Drug: Lidocaine 5% medicated Plaster
  Other Names: Versatis (Trade Mark); Lidoderm (Trade Mark); Neurodol Tissugel (Trade Mark)
  Arms: Lido-Patch (Double-blind Phase); Lido-Patch (Open-label Run-in Phase)
Drug: Placebo Plaster
  Arms: Placebo Patch (Double-blind Phase)

SUMMARY:
This study investigated the efficacy of the Lido-Patch (lidocaine 5% medicated plaster) in treatment of pain caused by PHN which is a neuropathic pain syndrome (nerve-related pain conditions) following an acute attack of herpes zoster (shingles).

DETAILED DESCRIPTION:
Participants were treated up to 10 weeks in this study: an 8-week Run-in Phase of open-label treatment with Lido-Patch was followed by a 2-day to 14-day Double-blind Phase with Lido-Patch or Placebo Patch treatment. Only participants responding to open-label treatment with Lido-Patch were included in the Double-blind Phase. In a Follow-up Phase without treatment, the safety of participants was monitored for 1-2 weeks. Alternatively, patch application could be continued for up to 12 months in the clinical study KF10004/02.

ELIGIBILITY:
Inclusion Criteria for the Run-in Phase:

* Adult participants, male and female, with a minimum age of 50 years at screening.
* Participants who had postherpetic neuralgia (PHN) for at least 3 months after healing of a herpes zoster skin rash.
* Pain score of at least 4, based on an 11-point numerical rating scale (NRS) (scale of 0-10), at the screening and enrolment visit. The pain assessment is the participant's recall of the pain intensity since the previous week.
* Written informed consent given.

Randomization Criteria:

* Participants must be regularly (minimum every second day) using the Lido-Patch for control of pain in the last 4 weeks of the run-in phase. The participant must wait for pain to increase before applying a new patch.
* The participants' average daily pain intensity (with patch on) must be 7 or less on an 11-point NRS (scale of 0-10), and must increase during the phases when a patch is not worn, during Week 8 of the Run-in Phase.
* Before randomization, the participant must have an average relief with Lido-Patch of "moderate" or better, on a 6-item scale (worse, no pain relief, slight, moderate, a lot, complete) during Week 8 of the Run-in Phase.

Exclusion Criteria:

* Participation in another study of investigational drugs or devices parallel to, or less than 30 days before screening, or previous participation in this study.
* Known to or suspected of not being able to comply with the study protocol.
* Any clinically significant condition that would, in the investigator's opinion, preclude study participation for instance alcohol, medication or drug dependency, neurotic personality, psychiatric illness, epilepsy or suicide risk.
* Pregnancy or nursing mother.
* Woman in childbearing age without satisfactory contraception.
* Hypersensitivity to lidocaine or amide-type local anesthetic drugs.
* Active herpes zoster lesion or dermatitis of any origin at the affected site with PHN.
* Evidence of another cause for pain in the area affected by herpes zoster in addition to PHN, such as lumbar radiculopathy, surgery or trauma, if this could confound assessment or self-evaluation of the pain due to post herpetic neuralgia.
* Participants who had neurological ablation by block or neurosurgical intervention for control of pain in PHN.
* Participants using topically applied analgesic compounds on the PHN affected area.
* Presence of other severe pain that could confound assessment or self-evaluation of the pain due to PHN.
* Participants with severe hepatic disorder and/or alanine or aspartate aminotransferase equal to or above 3-fold the upper limit of normal (ULN).
* Participants with severe renal disorder and/or increased serum creatinine equal to or above 1.5-fold the upper limit of normal (ULN).
* Participants who are undergoing active treatment for cancer, are known to be infected with the human immunodeficiency virus (HIV), or being acutely and intensively immunosuppressed following transplantation.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 265 (Actual)
Dates: Start 2003-04-29 (Actual); Primary Completion 2004-06-30 (Actual); Study Completion 2004-06-30 (Actual)

PRIMARY OUTCOMES:
Time-to-exit in Double-blind Phase Due to Lack of Efficacy | From Day 1 until time to exit in Double-blind Phase (maximum Day 14)
  The time to exit was defined as the number of days after randomization where worsening of the pain relief score by 2 or more categories on a 6-item pain relief scale (verbal rating scale, VRS) on 2 consecutive days in comparison to the average pain relief in Week 8 of the Run-in Phase was reported.
  The average pain relief in Week 8 of the enrichment phase was to be stated by the participant at the randomization visit. The VRS comprised the categories 1 = worse, 2 = no pain relief, 3 = slight, 4 = moderate, 5 = a lot, 6 = complete.

SECONDARY OUTCOMES:
Daily Pain Intensity: NRS | From screening visit (Week -1) to end of Double-blind Phase visit (Week 10)
  Pain intensity was assessed as "pain right now" directly before patch application and before patch removal, and as "24-hour average pain" before patch removal using an 11-point Numeric Rating Scale (NRS from 0 = no pain to 10 = pain as bad as you can imagine).
Daily Pain Relief | From screening visit (Week -1) to end of Double-blind Phase visit (Week 10)
  Pain relief was defined as relief at the time point directly before patch removal in comparison to the time point directly before patch application. Pain relief was assessed using a 6-item relief scale (VRS) with categories 1 = worse, 2 = no pain relief, 3 = slight, 4 = moderate, 5 = a lot, and 6 = complete.
Weekly Average 24-hour Pain Intensity: NRS | During Run-in Phase (visits after 1 and 4 weeks), after 8 weeks, and after 10 weeks (Double-blind Phase)
  The weekly average of the 24-hour average pain intensity was calculated based on corresponding daily pain intensities over the last week before the respective visit. Pain intensities were assessed using an 11-point Numeric Rating Scale (NRS from 0 = no pain to 10 = pain as bad as you can imagine).
Weekly Average Current Pain Intensity: NRS | During Run-in Phase (visits after 1 and 4 weeks), after 8 weeks, and after 10 weeks (Double-blind Phase)
  The weekly average of the current pain ("pain right now") intensities before patch application or before patch removal were calculated based on corresponding daily pain intensities over the last week before the respective visit. Pain intensities were assessed using an 11-point Numeric Rating Scale (NRS from 0 = no pain to 10 = pain as bad as you can imagine).
Weekly Average Pain Relief: VRS | During Run-in Phase (visits after 1 and 4 weeks), after 8 weeks, and after 10 weeks (Double-bind Phase)
  The weekly average pain relief was calculated based on daily pain relief over the last week before visit. Pain relief was assessed using a 6-item relief scale (VRS) with categories 1 = worse, 2 = no pain relief, 3 = slight, 4 = moderate, 5 = a lot, and 6 = complete.
Weekly Worst Pain Intensity: NRS | During Run-in Phase (visits after 1 and 4 weeks), after 8 weeks, and after 10 weeks (Double-blind Phase)
  Weekly worst pain intensity was assessed in the last week before the visit using an 11-point NRS (from 0 = no pain to 10 = pain as bad as you can imagine).
Weekly Average Pain Intensity: NRS | During Run-in Phase (visits after 1 and 4 weeks), after 8 weeks, and after 10 weeks (Double-blind Phase)
  Weekly average pain intensity was assessed in the last week before the visit using an 11-point NRS (from 0 = no pain to 10 = pain as bad as you can imagine).
Weekly Least Pain Intensity: NRS | During Run-in Phase (visits after 1 and 4 weeks), after 8 weeks, and after 10 weeks (Double-blind Phase)
  Weekly least pain intensity was assessed in the last week before the respective visit using an 11-point NRS (from 0 = no pain to 10 = pain as bad as you can imagine).

OTHER OUTCOMES:
Chronic Pain Sleep Inventory (CPSI) | From screening at each visit up to the final visit (Week 10) [6 time points in total]
  The CPSI is a 5-point verbal rating scale (VRS) designed to provide information on the influence of the pain on sleep quality with the items trouble falling asleep, needing sleep medication, and awakened by pain during the night/in the morning (categories of the VRS: never, rarely, sometimes, usually, always); in addition, the overall quality of sleep (categories of the VRS: poor, fair, good, very good, and excellent) was assessed. Participants were asked to complete the CPSI questionnaire at each visit.
Short Form McGill Pain Questionnaire (SF-MPQ) | At screening visit (Week -1), randomization visit (Week 8), and final visit (Week 10)
  The SF-MPQ includes 15 words (11 sensory, 4 affective). Each word or phrase is rated on a 4-point intensity scale (0 = none, 1 = mild, 2 = moderate, and 3 = severe). In addition, the 6-point Present Pain Intensity (PPI) rating (no pain, mild, discomforting, distressing, horrible, excruciating) is included as a visual analogue scale for rating pain intensity.
Clinical Global Impression of Change (CGIC) | Withdrawal visit (end of Run-in Phase) or final visit (end of Double-blind Phase)
  Investigators were to describe their global impression of change (CGIC), i.e., the overall impression of the change of the participant's condition by answering the question "Compared to the patient's condition at admission to the project, how much has he/she changed?" The verbal rating scale comprises the categories not assessed [0], very much improved [1], much improved [2], minimally improved [3], no change [4], minimally worse [5], much worse [6], and very much worse [7]. When assessing the overall impression, the investigator was to refer to the Run-in Phase only.
Short Form-36 Quality of Life Index (SF-36) | At screening visit (Week -1), randomization visit (Week 8), and final visit (Week 10)
  The Short Form 36 Quality of Life Index (SF-36 [Trade Mark]) standard version with a 4-week recall period was used as a self-assessment.
  Eleven questions were answered on binomial (Yes/No) or on 3-, 5-, or 6-point categorical scales to generate the 8 raw scales (Physical Functioning, Role-Physical, Bodily Pain, General Health, Vitality, Social Functioning, Role-Emotional, Mental Health). Higher values of the raw scales represent a better outcome. The raw scales were converted into a transformed scale (transformed scale = [(actual raw score - lowest possible raw score) / possible raw score range] x 100).
Allodynia Assessment | From screening at each visit up to Week 10 (6 time points in total)
  Allodynia severity was rated using the following categorical scale: 0 = no pain or discomfort to touch; 1 = uncomfortable, but tolerable to touch; 2 = painful; 3 = extremely painful, participant cannot stand touching.
  The test was conducted by means of a brush (type N12). The painful PHN area was stroked with the brush and the intensity of allodynic pain was assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Grünenthal Study Director, Study Director — Grünenthal GmbH

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Binder A, Bruxelle J, Rogers P, Hans G, Bosl I, Baron R. Topical 5% lidocaine (lignocaine) medicated plaster treatment for post-herpetic neuralgia: results of a double-blind, placebo-controlled, multinational efficacy and safety trial. Clin Drug Investig. 2009;29(6):393-408. doi: 10.2165/00044011-200929060-00003. PMID 19432499